CLINICAL TRIAL: NCT03276598
Title: A Randomised Double-blind Cross-over Single-centre Study on Molecular Genetics of Drug Responsiveness in Essential Hypertension
Brief Title: A Study on Molecular Genetics of Drug Responsiveness in Essential Hypertension
Acronym: GENRES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Kimmo Kontula, Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GENRES
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Hypertension; Pharmacogenetics
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Bisoprolol; Hydrochlorothiazide; Losartan

STUDY DESIGN:
Intervention Model Description: The design of the study is a randomized placebo-controlled cross-over study. The study starts with a run-in placebo period lasting for four weeks. The four monotherapy treatment periods last for four weeks and they are separated by placebo periods lasting also for four weeks. Randomization occurs after the first placebo period in blocks of 24 (all possible drug sequences).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo tablets and drugs are packed in similar gelatin capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Amlodipine (Active Comparator): One of the four monotherapy treatment periods.
  Interventions: Drug: Amlodipine
- Bisoprolol (Active Comparator): One of the four monotherapy treatment periods.
  Interventions: Drug: Bisoprolol
- Hydrochlorothiazide (Active Comparator): One of the four monotherapy treatment periods.
  Interventions: Drug: Hydrochlorothiazide
- Losartan (Active Comparator): One of the four monotherapy treatment periods.
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Placebo treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlodipine — Treatment for four weeks. Dose: 5 mg o.d.
  Arms: Amlodipine
Drug: Bisoprolol — Treatment for four weeks. Dose: 5 mg o.d.
  Arms: Bisoprolol
Drug: Hydrochlorothiazide — Treatment for four weeks. Dose: 25 mg o.d.
  Arms: Hydrochlorothiazide
Drug: Losartan — Treatment for four weeks. Dose: 50 mg o.d.
  Arms: Losartan
Drug: Placebo — Treatment for four weeks. Dose: 1 tablet per day.
  Arms: Placebo

SUMMARY:
Blood pressure variation and the risk of essential hypertension have an important genetic component. In most cases susceptibility to essential hypertension is likely determined by the action of more than one gene.

The identification of genes causing susceptibility to hypertension is important, since it would give new tools for the diagnosis and enable better etiological classification and specific treatment of the disease.

The innovation of this study is to use the response to antihypertensive therapy as an intermediate phenotype.

In the study, each subject uses one of four antihypertensive drugs, each as a monotherapy in a rotational fashion, for 28 days in a randomized order. The antihypertensive drugs to be tested include a thiazide diuretic, a beta-adrenergic antagonist, an angiotensin-II receptor antagonist and a calcium channel blocker. The drugs that are selected for the study are "typical" representatives of their groups and long-acting, and the dosages are sufficient but well tolerable.

DETAILED DESCRIPTION:
Blood pressure variation and the risk of essential hypertension have an important genetic component. In most cases susceptibility to essential hypertension is likely determined by the action of more than one gene.

The identification of genes causing susceptibility to hypertension is important, since it would give new tools for the diagnosis and enable better etiological classification and specific treatment of the disease. Finland is an ideal place for a study like this because of the genetic homogeneity of the population, the relatively high prevalence of the disease and the established protocols for the treatment and follow-up of hypertension in public health care.

The molecular genetic studies on hypertension performed so far (by 1999) have primarily been association studies, which are based on case-control classification and may produce erroneous results. Particularly, a reliable phenotyping of cases and controls has been difficult. Consequently, more attention should be paid to the phenotyping of patients, and novel intermediate phenotypes characteristic of certain subtypes of hypertension should be used to facilitate the search for hypertension genes. The innovation of this study is to use the response to antihypertensive therapy as an intermediate phenotype.

In the study, each subject uses one of four antihypertensive drugs, each as a monotherapy in a rotational fashion, for 28 days in a randomized order. The antihypertensive drugs to be tested include a thiazide diuretic, a beta-adrenergic antagonist, an angiotensin-II receptor antagonist and a calcium channel blocker. The drugs that are selected for the study are "typical" representatives of their groups and long-acting, and the dosages are sufficient but well tolerable. The study design does not necessitate the use of equipotent doses of the various agents, since the study is not designed to compare the antihypertensive effectiveness of the study drugs or, due to the short treatment periods, their effects on clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* essential hypertension diagnosed on an earlier occasion or during the present study (three diastolic blood pressure readings >=95 mmHg on separate occasions are required).

Exclusion Criteria (before and during the study):

* usage of three or more antihypertensive drugs
* secondary hypertension
* left ventricular hypertrophy
* drug-treated diabetes mellitus
* coronary heart disease
* stroke and other disorders of cerebral circulation
* renal disease
* obstructive pulmonary disease
* a disease treated with corticosteroids
* a disease with drug treatment potentially influencing blood pressure levels
* significant obesity (BMI >=32 kg/m2)
* allergic reaction towards any of the study drugs
* The patient is excluded from the study if his blood pressure level rises to 200/120 mmHg or above during the study.

Ages: 35 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 233 (Actual)
Dates: Start 1999-11-25 (Actual); Primary Completion 2004-04-01 (Actual); Study Completion 2004-04-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 4 weeks
  Change in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo K Kontula, Professor, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hiltunen TP, Suonsyrja T, Hannila-Handelberg T, Paavonen KJ, Miettinen HE, Strandberg T, Tikkanen I, Tilvis R, Pentikainen PJ, Virolainen J, Kontula K. Predictors of antihypertensive drug responses: initial data from a placebo-controlled, randomized, cross-over study with four antihypertensive drugs (The GENRES Study). Am J Hypertens. 2007 Mar;20(3):311-8. doi: 10.1016/j.amjhyper.2006.09.006. PMID 17324745
- [Result] Suonsyrja T, Hannila-Handelberg T, Paavonen KJ, Miettinen HE, Donner K, Strandberg T, Tikkanen I, Tilvis R, Pentikainen PJ, Kontula K, Hiltunen TP. Laboratory tests as predictors of the antihypertensive effects of amlodipine, bisoprolol, hydrochlorothiazide and losartan in men: results from the randomized, double-blind, crossover GENRES Study. J Hypertens. 2008 Jun;26(6):1250-6. doi: 10.1097/HJH.0b013e3282fcc37f. PMID 18475165
- [Result] Hiltunen TP, Donner KM, Sarin AP, Saarela J, Ripatti S, Chapman AB, Gums JG, Gong Y, Cooper-DeHoff RM, Frau F, Glorioso V, Zaninello R, Salvi E, Glorioso N, Boerwinkle E, Turner ST, Johnson JA, Kontula KK. Pharmacogenomics of hypertension: a genome-wide, placebo-controlled cross-over study, using four classes of antihypertensive drugs. J Am Heart Assoc. 2015 Jan 26;4(1):e001521. doi: 10.1161/JAHA.115.001778. PMID 25622599
- [Derived] Nuotio ML, Sanez Tahtisalo H, Lahtinen A, Donner K, Fyhrquist F, Perola M, Kontula KK, Hiltunen TP. Pharmacoepigenetics of hypertension: genome-wide methylation analysis of responsiveness to four classes of antihypertensive drugs using a double-blind crossover study design. Epigenetics. 2022 Nov;17(11):1432-1445. doi: 10.1080/15592294.2022.2038418. Epub 2022 Feb 25. PMID 35213289
- [Derived] Ala-Mutka EM, Rimpela JM, Fyhrquist F, Kontula KK, Hiltunen TP. Effect of hydrochlorothiazide on serum uric acid concentration: a genome-wide association study. Pharmacogenomics. 2018 Apr;19(6):517-527. doi: 10.2217/pgs-2017-0184. Epub 2018 Mar 27. PMID 29580174